CLINICAL TRIAL: NCT03079102
Title: Inhaled Nitric Oxide After Out-of-Hospital Cardiac Arrest
Acronym: iNOOHCA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment and planned change of institution by PI
Sponsor: Cameron Dezfulian (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Cameron Dezfulian, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO16100408
Record Dates: First submitted 2017-01-05; First posted 2017-03-14 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Heart Arrest, Out-Of-Hospital
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Nitric Oxide; Inosine; Endothelium-Dependent Relaxing Factors; Nitrogen

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to either placebo or active study drug (iNO). This will be stratified within blocks of 8 subjects at each center.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Gas canisters will be marked with a bar code which will be recorded by the study coordinator and available to the study team. Only the respiratory therapy directors will be aware of the canister content (placebo vs. active drug). Treatment assignment will be revealed upon opening a sealed opaque envelope after enrollment has been confirmed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- inhaled nitric oxide (iNO) (Experimental): 20 ppm iNO delivered via mechanical ventilator connected to the iNO ventilator delivery system (iNOvent). Drug will be started as soon as possible after return of spontaneous circulation (ROSC) but no later than 4h after ROSC. Study drug will be dosed for 12h then tapered off over 1h.
  Interventions: Drug: Nitric Oxide
- Placebo (Placebo Comparator): Nitrogen carrier gas delivered by identical system with similar dose/taper.
  Interventions: Drug: Nitrogen

INTERVENTIONS:
Drug: Nitric Oxide — An endogenous gaseous signaling molecule which stimulates soluble guanylate cyclase and may act via S-nitrosation, nitrite/nitrate or nitrated fatty acid formation.
  Other Names: inhaled nitric oxide, iNO, iNOMax
  Arms: inhaled nitric oxide (iNO)
Drug: Nitrogen — Nitrogen is the carrier gas (vehicle) for iNO. Subjects receiving placebo will receive equivalent doses of nitrogen.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Phase II double blind (participants and investigator) placebo controlled randomized (1:1) clinical trial of inhaled nitric oxide (iNO) 20 ppm administered over 12h beginning as soon as possible but within 4 h of return of spontaneous circulation (ROSC) from out-of-hospital cardiac arrest (OHCA). Planned enrollment is 180 subjects over 48 months at University of Pittsburgh Medical Center (UPMC) Hospitals with randomization stratified in blocks of 8. Recruitment will be performed under exception from informed consent (EFIC) to facilitate early enrollment and treatment. The study will have a pre-specified safety analysis at the mid-point (after 1 year or 60 patients whichever occurs first). Subjects will be screened by members of the University of Pittsburgh post-cardiac arrest service (PCAS), all of whom will serve as the study co-investigators, and the Research Coordinators. Notification of inclusion under EFIC will be performed as soon as possible by a member of the study team generally to a surrogate as the subjects will be comatose after OHCA.

DETAILED DESCRIPTION:
Subjects will be identified upon emergency department (ED) arrival or upon transfer from an outside facility and screened for enrollment by a PCAS physician as soon as possible. Eligible patients will have receive any required resuscitation (including central venous and arterial line placement, endotracheal intubation and hemodynamic resuscitation as needed) prior to having baseline labs and studies performed. Subjects will then be started on study drug delivered via the mechanical ventilator with a concealed canister (subject, providers and outcome assessors blind to treatment assignment). Randomization will be performed 1:1 in blocks of 8 using a random number generator. A randomization list will be prepared in advance by the director of respiratory therapy (RT) at each site and verified by a company representative. These individuals (who are not part of the study team) will be unblinded and assure that allocation to placebo and intervention is accurate. The allocation list will assign study drug canisters (by barcode) to each subject in order of study ID. Treatment assignment will be revealed after opening a sealed opaque envelope once enrollment is confirmed by a physician investigator. Study drug will then be administered by RT based on allocation. During study drug administration hourly vital signs will be obtained and methemoglobin levels for safety. Study drug will be weaned off after 12h over the course of 1h (10, 5, 4, 3, 2, 1 ppm each for 10 min) prior to discontinuation. Subjects will then receive standard post-resuscitation care with outcomes assessed by a blinded study team member (see below for outcomes).

Additional clinical variables to be collected Demographics and baseline function. Age, sex, race, maximum education level, employment status, marital status, Barthel activities of daily living (ADL) index prior to OHCA.

Arrest data. Location of OHCA, witnessed, bystander cardiopulmonary resuscitation (CPR), estimated no flow and low flow times, presenting rhythm, doses of epinephrine administered, shocks administered, recurrent arrest, date and time of ROSC.

Medical comorbidities. Diabetes, hypertension, active smoking, hyperlipidemia, chronic obstructive pulmonary disease (COPD), hypertension, drug abuse, prior myocardial infarction, prior coronary artery bypass grafting (CABG), prior coronary angiography with angioplasty or stent, congestive heart failure (EF on last echocardiogram [ECHO] prior to OHCA), obstructive sleep apnea, pulmonary hypertension, calculated Charlson comorbidity index (CCI).

Home medications. Statins, nitrates, anticoagulation, antiplatelet agents Hospital Interventions. Coronary angiography, percutaneous coronary intervention, CABG, mechanical ventilation hours and fraction of inspired oxygen (FiO2) from 0-24h after therapy start In-hospital medications. Alteplase, anti-epileptic medication use (valproate, phenytoin, lacosamide, levetiracetam), neurostimulants (methylphenidate, bromocriptine, modafinil, amantadine), cumulative dose of fentanyl, propofol, midazolam, cis-atracurium and vecuronium in at 24 (+/- 12 hours), 48 (+/- 12 hours), and 72 (+/- 12 hours) hours after therapy initiation

Data Storage Subjects will be assigned a study identifier (ID) upon entry and all data/samples stored using that ID. Linkage to patient identifiers will be maintained in a secure spreadsheet and will include name, date of birth and medical record number. Clinical data will be entered on case report forms (source documentation) which will be stored in a locked filing cabinet within a locked office assigned to the study team. Deidentified clinical and lab data will all be subsequently entered from the case report forms into a web based database (REDCap) to be maintained by Dr. Dezfulian's research assistant who has prior experience from other studies.

Statistical Analysis Plan Continuous data will be compared using t-tests and repeated measures ANOVA to compare between iNO and placebo groups at multiple times. Dichotomous outcomes including the primary endpoint will be compared by chi squared test. Time to awakening and 90d survival will be compared by log rank test of Kaplan-Meier survival plots. All tests will be two tailed with unadjusted p<0.05 considered significant. In the event of a differential distribution of baseline variables strongly associated with outcome (univariate OR >2), dichotomous outcomes will be adjusted for these baseline variables.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and comatose adult (>18 yo) resuscitated from out-of-hospital cardiac arrest (OHCA)*

  *Cardiac arrest within an emergency department or outpatient medical center will be included). OHCA includes Emergency Medical Service (EMS) witnessed cardiac arrest.
* Return of spontaneous circulation (ROSC) within 40 min of CPR initiation
* Full Outline of Unresponsiveness (FOUR) Brainstem score ≥ 2 (i.e. patient must have pupil OR corneal reflex at the time of ED presentation or within 1h if sedation/neuromuscular blockade clouds the picture)

Exclusion Criteria:

* Traumatic etiology of OHCA
* Prisoner
* Known pregnancy (beta-human chorionic gonadotropin screening is NOT REQUIRED for enrollment in women of appropriate age)
* Hemodynamic instability defined as >1 recurrent arrest prior to enrollment OR inability to maintain mean arterial blood pressure (MAP) > 65 using vasopressors and inotropes (ie actively up titrating medications or giving fluid bolus)
* Head CT grey-white ratio < 1.2; Head CT is NOT REQUIRED prior to enrollment
* Fixed and dilated pupils without another explanation
* Known intracranial hemorrhage or acute cerebral infarction; Head CT is NOT REQUIRED prior to enrollment
* Malignant EEG upon presentation defined as: myoclonic status epilepticus, non-convulsive status epilepticus, generalized periodic epileptiform discharges. EEG screening is NOT REQUIRED prior to enrollment
* ROSC >3h from time of ED arrival (treatment allocation must be within 4h so anything that will prevent this is reason for exclusion)
* Alert and interactive patient with minimal evidence of neurologic injury
* Plan to extubate within 12 hours
* Post-cardiac arrest service (PCAS) physician opinion that patient will die with >95% likelihood. This may be based on:

  * Multiple medical comorbidities
  * Late discovery of don not resuscitate (DNR) or advanced directive
  * Terminal diagnosis (other than OHCA; may have caused OHCA)
  * Clinical judgement based on current exam and data
* Patient is known to be taking phosphodiesterase type 5 (PDE5) inhibitors, soluble guanylyl cyclase (sGC) stimulator, or has a known diagnosis of Chronic thromboembolic pulmonary hypertension (CTEPH), pulmonary hypertension (PAH), or erectile dysfunction
* Known enrollment in another acute interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-08-26 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Dezfulian, MD, Principal Investigator — Assistant Professor of Critical Care Medicine and Clinical and Translational Science
Locations (5):
- United States (5):
  - UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC East, Monroeville, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magliocca A, Fries M. Inhaled gases as novel neuroprotective therapies in the postcardiac arrest period. Curr Opin Crit Care. 2021 Jun 1;27(3):255-260. doi: 10.1097/MCC.0000000000000820. PMID 33769417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were enrolled in the emergency room or intensive care unit. Screening for this study began on 8/21/2017. First enrollment was 8/26/2017 and the final enrollment was 4/25/2020.
Pre-assignment Details: Patients were assigned at the time of enrollment since enrollment was under exception from informed consent and all assigned patients were started on study drug.
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Started | 30 | 27
Completed | 30 | 26 (One subject had study drug discontinued by the PI after 3h of therapy due to progressive hemodynamic deterioration (worsening hypotension and shock). Discontinuation of study drug did not impact this deterioration.)
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [53 to 74] | 60 [44 to 72] | 64 [51.5 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 18 | 13 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 5 | 16
  White | 17 | 22 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 27 | 57
Height [Median (Inter-Quartile Range); unit: centimeters] | 171.5 [164 to 180] | 167.8 [160 to 175] | 170 [162.5 to 180]
Weight [Median (Inter-Quartile Range); unit: kilograms] | 86.6 [66.4 to 100] | 81.7 [69 to 111] | 85 [68.6 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death or Significant Neurological or Cardiac Impairment
Description: Composite of in-hospital death; OR unfavorable discharge location defined as a skilled nursing facility (SNF), long term acute care (LTAC) or hospice; OR New York Heart Association (NYHA) class III/IV heart failure at the time of discharge.*
  *In the setting of pre-existing heart failure there must be at least a 1 class decrement (eg III -> IV). If patient was previously housed in a "unfavorable" destination there must be a 1 point decrement (eg from SNF to LTAC or LTAC to hospice). Subjects with pre-existing NYHA IV symptoms or living in hospice are excluded from meeting the respective outcome.
Time Frame: Hospital discharge (+/- 3 days)
Population: All patients enrolled were followed to primary outcome consistent with FDA policies for trials conducted under exception from informed consent
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 30 | 27
Participants | 16 | 15

2. Secondary Outcome: Number of Subjects Dead
Description: Patient declared dead at designated time point
Time Frame: Hospital discharge (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 30 | 27
Participants | 13 | 11

3. Secondary Outcome: Number of Subjects Dead
Description: Patient declared dead at designated time point
Time Frame: 30 days after cardiac arrest (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 14 | 12

4. Secondary Outcome: Number of Subjects Dead
Description: Patient declared dead at designated time point
Time Frame: 90 days after cardiac arrest (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 27 | 25
Participants | 14 | 13

5. Secondary Outcome: Number of Subjects With a Favorable Cerebral Performance Category (CPC)
Description: The cerebral performance category (CPC) is a standardized scale from 1-5 describing neurological and functional outcome with a long history of use in cardiac arrest trials (N Engl J Med 1986; 314:397-403). Lower scores indicate better neurological performance as follows: (1) conscious and alert with normal function or only slight disability, (2) conscious and alert with moderate disability, (3) conscious with severe disability, (4) comatose or in a persistent vegetative state, or (5) dead. CPC will be dichotomized as favorable (1, 2) or unfavorable (3-5) at designated time.
Time Frame: Hospital discharge (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 30 | 27
Participants | 11 | 7

6. Secondary Outcome: Number of Subjects With a Favorable Cerebral Performance Category (CPC)
Description: as for outcome 5
Time Frame: 30 days after cardiac arrest (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 27 | 26
Participants | 8 | 9

7. Secondary Outcome: Number of Subjects With a Favorable Cerebral Performance Category (CPC)
Description: as for outcome 5
Time Frame: 90 days after cardiac arrest (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 27 | 27
Participants | 10 | 8

8. Secondary Outcome: Number of Subjects With a Favorable Modified Rankin Score (mRS)
Description: The modified Rankin Score (mRS) is now recommended by consensus as the best measure of neurologic outcome in cardiac arrest studies (Circulation. 2018;137:e783-e801). The mRS runs from 0-6, where higher numbers are consistent with more severe neurologic impairment up to death (6). The scores correspond to: (0) No symptoms; (1) No significant disability. Able to carry out all usual activities, despite some symptoms.;(2) Slight disability; (3) Moderate disability; (4) Moderately severe disability; (5) Severe disability; (6) Dead. This score was dichotomized as favorable (0-3) or unfavorable (4-6) at the appointed time.
Time Frame: Hospital discharge (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 30 | 27
Participants | 11 | 7

9. Secondary Outcome: Number of Subjects With a Favorable Modified Rankin Score (mRS)
Description: as for outcome 8
Time Frame: 30 days after cardiac arrest (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 27 | 26
Participants | 9 | 10

10. Secondary Outcome: Number of Subjects With a Favorable Modified Rankin Score (mRS)
Description: as for outcome 8
Time Frame: 90 days after cardiac arrest (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 27 | 23
Participants | 11 | 9

11. Secondary Outcome: Number of Subjects Discharged to a Favorable Destination
Description: Favorable discharge destination was defined as discharge from the hospital to home or inpatient rehabilitation. Unfavorable discharge destination was defined as discharge to a skilled nursing facility, long term acute care facility, hospice or death.
Time Frame: Hospital discharge (+/- 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 30 | 27
Participants | 15 | 12

12. Secondary Outcome: Barthel Index (Activities of Daily Living)
Description: Barthel Index of Independence in Activities of Daily Living scored as a continuous 0-100 at designated time. A higher score indicates improved ability to independently perform the activities of daily living.
Time Frame: Hospital discharge (+/- 3 days)
Population: One surviving subject in placebo group withdrew consent before discharge and was therefore not assessed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 17 | 15
score on a scale | 70 [30 to 100] | 65 [5 to 90]

13. Secondary Outcome: Barthel Index (Activities of Daily Living)
Description: as for outcome 12
Time Frame: 30 days after cardiac arrest (+/- 3 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 12 | 14
score on a scale | 100 [48.7 to 100] | 95 [3.75 to 100]

14. Secondary Outcome: Barthel Index (Activities of Daily Living)
Description: as for outcome 12
Time Frame: 90 days after cardiac arrest (+/- 3 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | 100 [100 to 100] | 100 [95 to 100]

15. Secondary Outcome: Time to Awakening
Description: Time in hours until subject is noted to follow commands. Subjects exceeding 96 hours of coma and those that die without awakening will be designated as 100.
Time Frame: Within 4 days of cardiac arrest
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 8 | 5
hours | 47.5 [25 to 100] | 25 [17 to 26]

16. Secondary Outcome: Methemoglobin Level
Description: Methemoglobin content as proportion (%) of total hemoglobin
Time Frame: Prior to study drug
Measure: Median (Inter-Quartile Range); unit: percentage of hemoglobin
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 6 | 4
percentage of hemoglobin | 0.1 [0 to 0.625] | 0.2 [0.1 to 0.4]

17. Secondary Outcome: Methemoglobin Level
Description: Methemoglobin content as proportion (%) of total hemoglobin
Time Frame: 6 hours after study drug initiated
Measure: Median (Inter-Quartile Range); unit: percentage of hemoglobin
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 17 | 14
percentage of hemoglobin | 1.1 [0.8 to 1.2] | 0.5 [0.4 to 0.6]

18. Secondary Outcome: Methemoglobin Level
Description: Methemoglobin content as proportion (%) of total hemoglobin
Time Frame: 12 hours after study drug initiated
Measure: Median (Inter-Quartile Range); unit: percentage of hemoglobin
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 6 | 6
percentage of hemoglobin | 0.8 [0.275 to 0.875] | 0.3 [0.125 to 0.55]

19. Secondary Outcome: Diastolic Blood Pressure
Description: Measured by arterial line
Time Frame: Hourly from 0 - 12 hours of study drug
Population: Missing values occurred due to death during study drug (iNO, 2; placebo, 1), withdrawal of consent (iNO, 1; placebo, 1), termination of study by PI and subsequent death (placebo, 1), procedures outside the ICU (placebo, 1), arterial line delay or malfunction (iNO, 1; placebo, 2).
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 29 | 26
mm Hg
  Time zero (immediately before study drug): number analyzed (Participants) | 28 | 23
  Time zero (immediately before study drug) | 75.1 (2.8) | 67.3 (3.7)
  1 hour after study drug: number analyzed (Participants) | 27 | 24
  1 hour after study drug | 72.5 (4.6) | 67.3 (2.2)
  2 hours after study drug: number analyzed (Participants) | 29 | 23
  2 hours after study drug | 72.1 (3.3) | 67.0 (4.2)
  3 hours after study drug: number analyzed (Participants) | 29 | 23
  3 hours after study drug | 71.3 (2.7) | 67.0 (2.3)
  4 hours after study drug: number analyzed (Participants) | 28 | 24
  4 hours after study drug | 71.6 (2.4) | 68.1 (3.6)
  5 hours after study drug: number analyzed (Participants) | 28 | 25
  5 hours after study drug | 72.6 (3.7) | 62.9 (2.2)
  6 hours after study drug: number analyzed (Participants) | 28 | 25
  6 hours after study drug | 74.9 (2.7) | 67.8 (3.1)
  7 hours after study drug: number analyzed (Participants) | 29 | 25
  7 hours after study drug | 68.7 (3.8) | 66.5 (4.1)
  8 hours after study drug: number analyzed (Participants) | 28 | 24
  8 hours after study drug | 71.5 (2.4) | 65.5 (3.5)
  9 hours after study drug: number analyzed (Participants) | 29 | 22
  9 hours after study drug | 70.8 (3.3) | 62.9 (2.3)
  10 hours after study drug: number analyzed (Participants) | 28 | 21
  10 hours after study drug | 71.4 (2.3) | 66.4 (3.7)
  11 hours after study drug: number analyzed (Participants) | 27 | 22
  11 hours after study drug | 70.7 (2.9) | 61.5 (2.0)
  12 hours after study drug: number analyzed (Participants) | 28 | 22
  12 hours after study drug | 67.0 (2.3) | 66.6 (3.2)

20. Secondary Outcome: Systolic Blood Pressure
Description: Measured by arterial line
Time Frame: Hourly from 0 - 12 hours of study drug
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 29 | 26
mm Hg
  0 hour (immediately before study drug start): number analyzed (Participants) | 28 | 23
  0 hour (immediately before study drug start) | 143.1 (6.6) | 140.0 (7.6)
  1 hour after study drug: number analyzed (Participants) | 27 | 24
  1 hour after study drug | 141.1 (6.6) | 136.1 (7.3)
  2 hours after study drug: number analyzed (Participants) | 29 | 23
  2 hours after study drug | 132.2 (5.2) | 140.5 (6.5)
  3 hours after study drug: number analyzed (Participants) | 29 | 23
  3 hours after study drug | 138.9 (5.3) | 132.5 (5.8)
  4 hours after study drug: number analyzed (Participants) | 28 | 24
  4 hours after study drug | 135.3 (4.5) | 134.3 (5.3)
  5 hours after study drug: number analyzed (Participants) | 28 | 25
  5 hours after study drug | 131.4 (3.9) | 134. (5.3)
  6 hours after study drug: number analyzed (Participants) | 28 | 25
  6 hours after study drug | 126.2 (4.0) | 139.8 (5.9)
  7 hours after study drug: number analyzed (Participants) | 29 | 25
  7 hours after study drug | 129.0 (3.8) | 128.8 (6.1)
  8 hours after study drug: number analyzed (Participants) | 28 | 24
  8 hours after study drug | 126.0 (4.0) | 132.2 (6.0)
  9 hours after study drug: number analyzed (Participants) | 29 | 22
  9 hours after study drug | 125.9 (3.9) | 132.5 (6.2)
  10 hours after study drug: number analyzed (Participants) | 28 | 21
  10 hours after study drug | 127.1 (3.8) | 136.8 (5.9)
  11 hours after study drug: number analyzed (Participants) | 27 | 22
  11 hours after study drug | 119.4 (3.7) | 136.7 (5.0)
  12 hours after study drug: number analyzed (Participants) | 28 | 22
  12 hours after study drug | 119.4 (3.7) | 134.2 (6.3)

21. Secondary Outcome: Heart Rate
Description: Calculated from continuous telemetry by monitor
Time Frame: Hourly from 0 - 12 hours of study drug
Population: Missing values occurred due to death during study drug (iNO, 2; placebo, 1), withdrawal of consent (iNO, 1; placebo, 1), termination of study by PI (placebo, 1), procedures outside the ICU (placebo, 1).
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 29 | 26
beats per minute
  0 hour (immediately before study drug) | 90.0 (3.8) | 31.1 (3.4)
  1 hour after study drug start | 85.2 (3.6) | 91.8 (5.5)
  2 hours after study drug start | 84.4 (3.2) | 85.7 (4.5)
  3 hours after study drug start: number analyzed (Participants) | 29 | 25
  3 hours after study drug start | 82.3 (3.3) | 85.9 (4.6)
  4 hours after study drug start: number analyzed (Participants) | 28 | 25
  4 hours after study drug start | 77.1 (3.0) | 83.6 (4.3)
  5 hours after study drug start: number analyzed (Participants) | 28 | 25
  5 hours after study drug start | 78.0 (2.9) | 79.8 (4.2)
  6 hours after study drug start: number analyzed (Participants) | 28 | 25
  6 hours after study drug start | 76.7 (3.1) | 77.5 (4.0)
  7 hours after study drug start: number analyzed (Participants) | 28 | 25
  7 hours after study drug start | 76.8 (3.3) | 74.9 (3.5)
  8 hours after study drug start: number analyzed (Participants) | 28 | 25
  8 hours after study drug start | 76.1 (3.9) | 76.0 (3.6)
  9 hours after study drug start: number analyzed (Participants) | 28 | 23
  9 hours after study drug start | 75.9 (4.0) | 75.0 (3.9)
  10 hours after study drug start: number analyzed (Participants) | 28 | 23
  10 hours after study drug start | 74.7 (3.9) | 75.4 (3.2)
  11 hours after study drug start: number analyzed (Participants) | 27 | 23
  11 hours after study drug start | 72.9 (3.8) | 75.7 (3.5)
  12 hours after study drug start: number analyzed (Participants) | 27 | 23
  12 hours after study drug start | 73.4 (3.5) | 75.9 (4.1)

ADVERSE EVENTS:
Time Frame: From start of study drug through hospital discharge, up to 90 days follow-up
Description: Common expected serious adverse events (SAEs) are listed below and defined:
  * Hypotension: systolic blood pressure ≤ 90 mmHg or mean arterial blood pressure ≤65 mmHg
  * Hypoxia: Arterial partial pressure oxygen (paO2) < 8 kPa (60 mmHg) when breathing room air or an oxygenation index (paO2:fraction of inspired oxygen [FiO2] ≤ 200 mmHg)
  * Metabolic acidosis: Arterial blood gas base deficit ≥ 5.0 mmol/L or serum lactate ≥ 3.6 mg/dL
  * Methemoglobin level > 10%
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
All-Cause Mortality (participants affected / at risk) | 14/30 | 13/27
Serious Adverse Events (participants affected / at risk) | 24/30 | 25/27
Other Adverse Events (participants affected / at risk) | 0/30 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Nitric Oxide (iNO) (N=30) | Placebo (N=27)
Hypotension (Cardiac disorders) | 10 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14 | 17
Metabolic acidosis (Metabolism and nutrition disorders) | 20 | 24
Methemoglobinemia (Blood and lymphatic system disorders) | 0 | 0 — Methemoglobin > 10%
Cardiac arrest (Cardiac disorders) | 0 | 4
Cerebral edema (Nervous system disorders) | 2 | 0
Stroke (Nervous system disorders) | 2 | 0
Myoclonic status epilepticus (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Planned Echocardiogram data was not able to be collected due to technical and feasibility constraints.

Laser speckle contrast imaging data still requires validation and is therefore not reported.

CPC-extended data was incomplete across many domains and therefore is not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT03079102/Prot_SAP_000.pdf